CLINICAL TRIAL: NCT06298513
Title: Autonomic and Metabolic Response to Cardiac Rehabilitation After Acute Myocardial Infarction
Brief Title: Autonomic and Metabolic Response to Cardiac Rehabilitation After Acute MI
Acronym: RIABILITOMICA
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 09C338
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Acute Myocardial Infarction: Rehabilitation Phase
Keywords: myocardial infarction; cardiac rehabilitation; metabolomic; autonomic nervous ststem
MeSH Terms: conditions — Myocardial Infarction | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — frozen plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient after first acute myocardial infarction
  Interventions: Other: Cardiac rehabilitation

INTERVENTIONS:
Other: Cardiac rehabilitation — Six weeks of cardiac rehabilitation with physical training

SUMMARY:
Ischemic heart disease remains the leading cause of death in the western world. The beneficial effects of cardiac rehabilitation on the evolution of ischemic heart disease are known, but the effects of rehabilitation on the metabolic processes of the patients are so far poorly understood. Metabolomics is the qualitative/quantitative analysis of the body's metabolic responses to pathophysiological stimuli or genetic alterations. Metabolic changes caused by physical activity have been demonstrated in obese and diabetic patients and in athletes. Aim of the study is to evaluate whether cardiac rehabilitation after a first myocardial infarction induces changes in the metabolic state of patients, and whether these changes may be related with changes in the usual risk factors (i.e. glyco-lipidic profile, natriuretic peptides, homocysteine).

ELIGIBILITY:
Inclusion Criteria:

* recent first acute myocardial infarction

Exclusion Criteria:

* severe diabetes

Ages: 25 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients meeting the eligibility criteria will be proposed to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Changes in purine after rehabilitation | Baseline and after 6 weeks of rehabilitation
  The concentration of purine will be calculated after rehabilitation, and compared to its baseline concentration by a paired T test analysis.
Changes in histidine after rehabilitation | Baseline and after 6 weeks of rehabilitation
  The concentration of purine will be calculated after rehabilitation, and compared to its baseline concentration by a paired T test analysis
Changes in galactose after rehabilitation | Baseline and after 6 weeks of rehabilitation
  The concentration of galactose will be calculated after rehabilitation, and compared to its baseline concentration by a paired T test analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy